CLINICAL TRIAL: NCT02782949
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Meriva® (Curcuminoids) as a Candidate Chemoprevention Agent for Gastric Carcinogenesis
Brief Title: Curcumin in Preventing Gastric Cancer in Patients With Chronic Atrophic Gastritis or Gastric Intestinal Metaplasia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2016-00713; NCI-2016-00713 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00042; MAY2015-05-01 (Other: Mayo Clinic in Rochester); MAY2015-05-01 (Other: DCP); N01CN00042 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2016-05-25; First posted 2016-05-26 (Estimated); Results first posted 2024-03-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Atrophic Gastritis; Gastric Carcinoma
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (curcumin) (Experimental): Patients receive curcumin PO BID for 180 days in the absence of unacceptable toxicity.
  Interventions: Drug: Curcumin; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for 180 days in the absence of unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Curcumin — Given PO
  Other Names: C.I. 75300; C.I. Natural Yellow 3; Diferuloylmethane; Turmeric Yellow
  Arms: Arm I (curcumin)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase IIb trial studies how well curcumin works in preventing gastric cancer in patients with chronic atrophic gastritis and/or gastric intestinal metaplasia. Curcumin is an antioxidant compound found in plants that may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the change in gastric mucosal interleukin 1beta (IL-1beta) cytokine level, quantified by Luminex assay technology, after a 6-month intervention in participants randomly assigned to the curcumin (Meriva [curcuminoids]) versus placebo arms.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of Meriva versus placebo. II. To compare changes in Histology Gastric Score (HGS) from baseline to 6 months for Meriva versus placebo.

III. To compare changes in additional gastric mucosal cytokine/chemokine levels (interleukin 8 [IL-8], tumor necrosis factor-alpha [TNFalpha], and inducible protein 10 [IP-10]; quantified by Luminex assay).

IV. To compare changes in gastric mucosal deoxyribonucleic acid (DNA) damage as assessed by immunohistochemistry (IHC), of the biomarkers 8-hydroxy-2'-deoxyguanosine (8-OHdG) and phosphorylated subtype of histone H2A (H2AX).

V. To explore associations between proinflammatory cytokine genotype status (IL-1beta, IL-8, and TNFalpha single nucleotide polymorphisms [SNPs]; characterized at baseline) and the above outcomes.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM 1: Patients receive curcumin orally (PO) twice daily (BID) for 180 days in the absence of unacceptable toxicity.

ARM 2: Patients receive placebo PO BID for 180 days in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and 7 months.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION CRITERIA
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to undergo screening tests and procedures
* Willingness to provide blood and tissue samples for safety/toxicity monitoring and biomarker analyses
* Willingness to avoid the use of curcumin or any over-the-counter or prescription medications containing curcumin or curcuminoids
* REGISTRATION/RANDOMIZATION INCLUSION CRITERIA
* Histologically-confirmed chronic multifocal atrophic gastritis (MAG) and/or gastric intestinal metaplasia (GIM)
* Helicobacter pylori negative, defined as negative stool antigen testing and negative histological examination
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Aspartate transaminase (AST), alanine transferase (ALT) within institutional limits of normal or judged to be not clinically significant by the investigator
* Alkaline phosphatase within institutional limits of normal or judged to be not clinically significant by the investigator
* Platelets within institutional limits of normal or judged to be not clinically significant by the investigator
* Hemoglobin within institutional limits of normal or judged to be not clinically significant by the investigator
* White blood cells (WBC) within institutional limits of normal or judged to be not clinically significant by the investigator
* Blood urea nitrogen (BUN) within institutional limits of normal or judged to be not clinically significant by the investigator
* Total bilirubin within institutional limits of normal or judged to be not clinically significant by the investigator
* Creatinine within institutional limits of normal or judged to be not clinically significant by the investigator
* Not pregnant or breast feeding; Note: The effects of Meriva on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, individuals of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION CRITERIA
* History of other malignancy =< 2 years prior to the registration/randomization evaluation, with the exception of basal cell or squamous cell skin cancer
* History of colorectal cancer; exception: individuals with stage I or II colorectal cancer who have not received any chemotherapy
* Known diagnosis of human immunodeficiency virus (HIV); Note: An HIV screening test does not have to be performed to evaluate this criterion
* History of gastric surgery
* Receiving any other investigational agents
* Use of any anticoagulation medications, such as warfarin or Coumadin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding; Note: Pregnant women are excluded from this study; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Meriva, breastfeeding should be discontinued if the mother is treated with Meriva
* REGISTRATION/RANDOMIZATION EXCLUSION CRITERIA
* Receiving any other investigational, anticoagulation, and/or chemotherapy agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Meriva

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2026-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia R Cruz-Correa, Principal Investigator — Mayo Clinic
Locations (2):
- Hospital Regional de Occidente, Santa Rosa de Copán, Honduras
- University of Puerto Rico, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Curcumin): Patients receive curcumin PO BID for 180 days in the absence of unacceptable toxicity.>
  > Curcumin: Given PO>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Quality-of-Life Assessment: Ancillary studies
- Arm II (Placebo): Patients receive placebo PO BID for 180 days in the absence of unacceptable toxicity.>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Placebo Administration: Given PO>
  > Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Started | 24 | 26
Completed | 23 | 25
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Curcumin): Patients receive curcumin PO BID for 180 days in the absence of unacceptable toxicity.
  >
  > Curcumin: Given PO
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Quality-of-Life Assessment: Ancillary studies
- Arm II (Placebo): Patients receive placebo PO BID for 180 days in the absence of unacceptable toxicity.
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Placebo Administration: Given PO
  >
  > Quality-of-Life Assessment: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Arm I (Curcumin) | Arm II (Placebo) | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (10.51) | 60.4 (10.77) | 61.2 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 48
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 13 | 24
  More than one race | 10 | 12 | 22
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Honduras | 10 | 12 | 22
  Puerto Rico | 14 | 14 | 28
Gastric mucosal histologic diagnosis [Count of Participants; unit: Participants]
  MAG (multifocal atrophic gastritis) | 5 | 6 | 11
  GIM (gastric intestinal metaplasia) | 16 | 17 | 33
  Both (from screening endoscopic gastroduodenoscopy or EGD) | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in IL-1beta Cytokine Levels in the Gastric Mucosa
Description: Will be measured by Luminex assay. If the data are not normally distributed, the Wilcoxon Rank-Sum test will be used. The 95% confidence intervals will also be provided.
Time Frame: Baseline up to 6 months
Population: Only 47 evaluable participants.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 22 | 25
pg/mL
  Antrum: IL-1beta Difference | 0.0 [-4.2 to 10.9] | -0.1 [-5.5 to 4.1]
  Body: IL-1beta Difference | 0.0 [-5.2 to 4.2] | 0.1 [-0.8 to 8.6]
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.3990, Wilcoxon Rank-Sum test

2. Secondary Outcome: Change in Histology Gastric Score
Description: Will compare changes in histology gastric score for curcumin versus placebo.
  Correa Histopathology Scoring System values according to the histological diagnosis categories Histological diagnosis Correa Histopathology Scores (range)
  1. Normal 1
  2. non-atrophic gastritis(NAG) 2
  3. multifocal atrophic gastritis without intestinal metaplasia (MAG) 3.25-4.00*
  4. IM (intestinal metaplasia) 4.30-5.00*
  5. Dysplasia 5.25-5.75*
  6. Gastric Cancer 6
Time Frame: Baseline up to 6 months
Population: Same populations. A central pathology review of pre-and post-intervention biopsy specimens was performed at the University of Puerto Rico for all study endpoints. Only 47 evaluable participants.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 22 | 25
scores on a scale
  Correa Score Difference (Puerto Rico data) central review | 0.0 [-2.8 to 3.6] | 0.0 [-3.6 to 2.6]
  Correa Score Difference (UAB data) | 0.0 [-3.6 to 3.6] | 0.0 [-3.9 to 3.5]

3. Secondary Outcome: Additional Gastric Mucosal Cytokine/Chemokine Levels (TNFalpha, and IP-10)
Description: Will be quantified with Luminex assay. Changes in the concentrations (or categories) will be explored within and between the intervention arms. Fisher's exact tests, Wilcoxon rank sum tests, and two-sample t-tests will be used to assess differences between groups. McNemar's tests, Wilcoxon signed rank tests, and paired sample t-tests will be used to assess differences within each arm. Graphical methods (i.e. boxplots, scatter plots, etc.) will also be used to describe the data.
Time Frame: Baseline up to 6 months
Population: Only 47 evaluable participants.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 22 | 25
pg/mL
  Antrum: TNF-alpha Difference | -0.1 [-3.8 to 5.7] | 0.0 [-1.8 to 8.7]
  Antrum: IP-10 Difference | 8.0 [-135.7 to 285.9] | 14.3 [-218.3 to 179.2]
  Body: IP-10 Difference | 1.2 [-356.5 to 217.0] | 5.2 [-132.3 to 157.9]
  Body: TNF-alpha Difference | 0.0 [-1.8 to 4.6] | 0.0 [-8.0 to 12.0]
  Antrum: IL-8 Difference | -0.3 [-30.7 to 12.4] | -0.2 [-55.4 to 385.2]
  Body: IL-8 Difference | 0.0 [-1.8 to 4.6] | 0.0 [-8.0 to 12.0]

4. Secondary Outcome: Gastric Mucosal Deoxyribonucleic Acid (DNA) Damage
Description: Will be assessed by immunohistochemistry. Fisher's exact tests, Wilcoxon rank sum tests, and two-sample t-tests will be used to assess differences between groups. McNemar's tests, Wilcoxon signed rank tests, and paired sample t-tests will be used to assess differences within each arm. Graphical methods (i.e. boxplots, scatter plots, etc.) will also be used to describe the data.
Time Frame: Baseline up to 6 months
Population: Only 47 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 22 | 25
Participants
  DNA Damage: Baseline: < 1% | 18 | 19
  DNA Damage: Baseline: 1-5% | 2 | 4
  DNA Damage: Baseline: >5% | 2 | 1
  DNA Damage: Baseline: Missing | 0 | 1
  DNA Damage: Month 6: < 1% | 19 | 13
  DNA Damage: Month 6: 1-5% | 2 | 10
  DNA Damage: Month 6: >5% | 1 | 1
  DNA Damage: Month 6: Missing | 0 | 1
Statistical Analysis 1: Comparison: Arm I (Curcumin) vs Arm II (Placebo); Test type: Superiority; p = 0.74, Fisher Exact

5. Other Pre Specified Outcome: Proinflammatory Cytokine Genotype Status (IL-1beta, IL-8, and TNFalpha Single Nucleotide Polymorphisms)
Description: Will be examined in relation to the outcomes above to further characterize the at-risk population and generate hypotheses for future studies.
Time Frame: At baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 7 months
Arm/Group | Arm II (Placebo) | Arm I (Curcumin)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 14/26 | 12/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm II (Placebo) (N=26) | Arm I (Curcumin) (N=24)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 2 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 2 (2) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT02782949/Prot_SAP_ICF_001.pdf